CLINICAL TRIAL: NCT02523911
Title: Sodium Sulfate/Potassium Sulfate/Magnesium Sulfate Bowel Preparation With and Without Simethicone for Routine Colonoscopy: A Double-blinded Randomized Controlled Trial
Brief Title: Efficacy and Tolerability of Suprep With and Without Simethicone for Routine Colonoscopy for Colorectal Cancer Screening
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator graduated and is not longer at this institution
Sponsor: MercyOne Des Moines Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: MMC2015-31
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer
Keywords: Suprep; Simethicone; Colorectal cancer screening; Routine colonoscopy; sodium sulfate/potassium sulfate/magnesium sulfate; Bowel cleansing; Mass screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Simethicone; sodium sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simethicone Group (Active Comparator): Early in the evening prior to colonoscopy, patients will be instructed to consume one 6 ounce bottle of oral sodium sulfate/potassium sulfate/magnesium sulfate (Suprep) solution (containing sodium sulfate 17.5 grams, potassium sulfate 3.13 grams, and magnesium sulfate 1.6 grams) diluted with 16 ounces of water over one hour. Over the next hour, the patient will be instructed to drink an additional 32 ounces of water. On the day of colonoscopy, the same procedure will be repeated. Patients will take 2.4 mL simethicone in a half glass of water immediately after consuming each dose of the Suprep. All of the bowel preparation solution and required water should be consumed at least 2 hours prior to colonoscopy.
  Interventions: Drug: Simethicone; Drug: sodium sulfate/potassium sulfate/magnesium sulfate solution
- Placebo Group (Placebo Comparator): Early in the evening prior to colonoscopy, patients will be instructed to consume one 6 ounce bottle of oral sodium sulfate/potassium sulfate/magnesium sulfate (Suprep) solution (containing sodium sulfate 17.5 grams, potassium sulfate 3.13 grams, and magnesium sulfate 1.6 grams) diluted with 16 ounces of water over one hour. Over the next hour, the patient will be instructed to drink an additional 32 ounces of water. On the day of colonoscopy, the same procedure will be repeated. Patients will take 2.4 mL of placebo (identical in appearance to simethicone) in a half glass of water immediately after consuming each dose of the Suprep. All of the bowel preparation solution and required water should be consumed at least 2 hours prior to colonoscopy.
  Interventions: Drug: Placebo; Drug: sodium sulfate/potassium sulfate/magnesium sulfate solution

INTERVENTIONS:
Drug: Simethicone — Patients will be randomized to receive either simethicone or placebo in addition to oral sodium sulfate/potassium sulfate/magnesium sulfate solution (Suprep), and will be blinded to whether they are in the simethicone arm or the placebo arm of the trial. Simethicone and placebo will be prepared as identically-appearing liquid solution (2.4 mL) with the assistance of a pharmacist. The simethicone or placebo solution will then be assigned to patients according to the randomization scheme and samples will be labeled with patient information prior to distribution. Only the pharmacist will participate in the labeling process and know which patients receive simethicone or placebo; administering staff, nurses, physicians, and patients will be blinded to this.
  Other Names: Gas-X Infant Drops; Infants Gas Relief; Infants Simethicone; Infants' Mylicon
  Arms: Simethicone Group
Drug: Placebo — Patients will be randomized to receive either simethicone or placebo in addition to oral sodium sulfate/potassium sulfate/magnesium sulfate solution (Suprep), and will be blinded to whether they are in the simethicone arm or the placebo arm of the trial. Simethicone and placebo will be prepared as identically-appearing liquid solution (2.4 mL) with the assistance of a pharmacist. The simethicone or placebo solution will then be assigned to patients according to the randomization scheme and samples will be labeled with patient information prior to distribution. Only the pharmacist will participate in the labeling process and know which patients receive simethicone or placebo; administering staff, nurses, physicians, and patients will be blinded to this.
  Other Names: Inert solution
  Arms: Placebo Group
Drug: sodium sulfate/potassium sulfate/magnesium sulfate solution — Both arms will receive sodium sulfate/potassium sulfate/magnesium sulfate solution for bowel preparation
  Other Names: Suprep Bowel Prep Kit

SUMMARY:
The purpose of this study is to investigate Suprep bowel preparation, with and without the anti-gas medication simethicone, in terms of efficacy and patient tolerability in the preparation of patients undergoing routine colonoscopy for colorectal cancer screening.

DETAILED DESCRIPTION:
The study will investigate sodium sulfate/potassium sulfate/magnesium sulfate (Suprep), with and without simethicone, in terms of efficacy and patient tolerability in the preparation of patients undergoing routine colonoscopy. Adult ambulatory outpatients who are scheduled for elective routine colonoscopy for colorectal cancer screening will be recruited to participate in the trial. Patients will be randomized to receive either simethicone or placebo in addition to oral sodium sulfate/potassium sulfate/magnesium sulfate solution (Suprep) and will receive verbal and written instruction on administration of solutions. During colonoscopy, three areas of the colon (right colon, transverse colon, and left colon) will be assessed during removal of the colonoscope for overall colon cleansing, presence of bubbles, and degree of haziness; this will be scored by a blinded endoscopist. A separate written patient questionnaire will be used to assess acceptability and tolerability of the preparation, as well as any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Outpatients who require elective colonoscopy for colorectal cancer screening at Iowa Endoscopy Center and at University of Florida - Jacksonville

Exclusion Criteria:

* Allergy or hypersensitivity to any constituent of the lavage solution or to simethicone
* Presence of any contraindication to colonoscopy (i.e. uncontrolled congestive heart failure, New York Heart Association classification III-IV, history of myocardial infarction within 6 months, coagulopathy)
* Massive ascites
* Renal insufficiency
* Pregnancy
* History of colonic surgery
* History of anti-flatulence or laxative agent within one week
* Refusal/inability to give consent
* Patients undergoing colonoscopy for reasons other than colorectal cancer screening
* Mentally disabled
* Non-English-speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall bowel cleansing | During procedure
  To be assessed during removal of the colonoscope during the procedure and blinded endoscopist will score using a written questionnaire

SECONDARY OUTCOMES:
Number of patients with adverse effects | Day prior to and day of colonoscopy
  A written patient questionnaire will be used to assess patient acceptability and tolerability by recording any adverse effects experienced, including nausea, vomiting, headache, insomnia, bloating, abdominal pain, abdominal discomfort, abdominal cramps or any others.
Number of patients completing the bowel preparation | Day prior to and day of colonoscopy
  A written patient questionnaire will be used to assess compliance by asking if the total prescribed volume of solution was ingested and by recording number of evacuations.

OTHER OUTCOMES:
Presence of bubbles | During procedure
  To be assessed during removal of the colonoscope during the procedure and blinded endoscopist will score using a written questionnaire
Degree of haziness | During procedure
  To be assessed during removal of the colonoscope during the procedure and blinded endoscopist will score using a written questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tercio Lopes, MD, Principal Investigator — Iowa Digestive Disease Center; Silvio de Melo, MD, Principal Investigator — University of Florida Health Systems, Jacksonville
Locations (2):
- United States (2):
  - UF Health Jacksonville, Jacksonville, Florida
  - Iowa Endoscopy Center, Clive, Iowa

REFERENCES:
- [Background] Valiante F, Bellumat A, De Bona M, De Boni M. Bisacodyl plus split 2-L polyethylene glycol-citrate-simethicone improves quality of bowel preparation before screening colonoscopy. World J Gastroenterol. 2013 Sep 7;19(33):5493-9. doi: 10.3748/wjg.v19.i33.5493. PMID 24023492
- [Background] Gentile M, De Rosa M, Cestaro G, Forestieri P. 2 L PEG plus ascorbic acid versus 4 L PEG plus simethicon for colonoscopy preparation: a randomized single-blind clinical trial. Surg Laparosc Endosc Percutan Tech. 2013 Jun;23(3):276-80. doi: 10.1097/SLE.0b013e31828e389d. PMID 23751992
- [Background] Pontone S, Angelini R, Standoli M, Patrizi G, Culasso F, Pontone P, Redler A. Low-volume plus ascorbic acid vs high-volume plus simethicone bowel preparation before colonoscopy. World J Gastroenterol. 2011 Nov 14;17(42):4689-95. doi: 10.3748/wjg.v17.i42.4689. PMID 22180711
- [Background] Jansen SV, Goedhard JG, Winkens B, van Deursen CT. Preparation before colonoscopy: a randomized controlled trial comparing different regimes. Eur J Gastroenterol Hepatol. 2011 Oct;23(10):897-902. doi: 10.1097/MEG.0b013e32834a3444. PMID 21900786
- [Background] Park JJ, Lee SK, Jang JY, Kim HJ, Kim NH. The effectiveness of simethicone in improving visibility during colonoscopy. Hepatogastroenterology. 2009 Sep-Oct;56(94-95):1321-5. PMID 19950784
- [Background] Tongprasert S, Sobhonslidsuk A, Rattanasiri S. Improving quality of colonoscopy by adding simethicone to sodium phosphate bowel preparation. World J Gastroenterol. 2009 Jun 28;15(24):3032-7. doi: 10.3748/wjg.15.3032. PMID 19554657
- [Background] Sudduth RH, DeAngelis S, Sherman KE, McNally PR. The effectiveness of simethicone in improving visibility during colonoscopy when given with a sodium phosphate solution: a double-bind randomized study. Gastrointest Endosc. 1995 Nov;42(5):413-5. doi: 10.1016/s0016-5107(95)70041-2. PMID 8566629
- [Background] Lazzaroni M, Petrillo M, Desideri S, Bianchi Porro G. Efficacy and tolerability of polyethylene glycol-electrolyte lavage solution with and without simethicone in the preparation of patients with inflammatory bowel disease for colonoscopy. Aliment Pharmacol Ther. 1993 Dec;7(6):655-9. doi: 10.1111/j.1365-2036.1993.tb00148.x. PMID 8161673
- [Background] Shaver WA, Storms P, Peterson WL. Improvement of oral colonic lavage with supplemental simethicone. Dig Dis Sci. 1988 Feb;33(2):185-8. doi: 10.1007/BF01535731. PMID 3338367
- [Background] Wexner SD, Beck DE, Baron TH, Fanelli RD, Hyman N, Shen B, Wasco KE; American Society of Colon and Rectal Surgeons; American Society for Gastrointestinal Endoscopy; Society of American Gastrointestinal and Endoscopic Surgeons. A consensus document on bowel preparation before colonoscopy: prepared by a task force from the American Society of Colon and Rectal Surgeons (ASCRS), the American Society for Gastrointestinal Endoscopy (ASGE), and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Gastrointest Endosc. 2006 Jun;63(7):894-909. doi: 10.1016/j.gie.2006.03.918. No abstract available. PMID 16733101
- [Background] Chiu HM, Lin JT, Wang HP, Lee YC, Wu MS. The impact of colon preparation timing on colonoscopic detection of colorectal neoplasms--a prospective endoscopist-blinded randomized trial. Am J Gastroenterol. 2006 Dec;101(12):2719-25. doi: 10.1111/j.1572-0241.2006.00868.x. Epub 2006 Oct 6. PMID 17026559
- [Background] McNally PR, Maydonovitch CL, Wong RK. The effect of simethicone on colonic visibility after night-prior colonic lavage. A double-blind randomized study. J Clin Gastroenterol. 1989 Dec;11(6):650-2. doi: 10.1097/00004836-198912000-00010. PMID 2584664
- [Background] McNally PR, Maydonovitch CL, Wong RK. The effectiveness of simethicone in improving visibility during colonoscopy: a double-blind randomized study. Gastrointest Endosc. 1988 May-Jun;34(3):255-8. doi: 10.1016/s0016-5107(88)71324-3. PMID 3292345
- [Background] Wu L, Cao Y, Liao C, Huang J, Gao F. Systematic review and meta-analysis of randomized controlled trials of Simethicone for gastrointestinal endoscopic visibility. Scand J Gastroenterol. 2011 Feb;46(2):227-35. doi: 10.3109/00365521.2010.525714. Epub 2010 Oct 26. PMID 20977386